CLINICAL TRIAL: NCT06819813
Title: Open Trial of a Technology-Based Intervention for Dysregulated Eating in Adolescents With or At Risk for Overweight or Obesity
Brief Title: Project VIBE: Virtual Intervention for Binge Eating in Adolescents
Acronym: VIBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Northwestern University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andrea Goldschmidt, Associate Professor of Psychiatry, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23020100; R01DK136540-01 (NIH)
Record Dates: First submitted 2025-01-28; First posted 2025-02-11 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Binge-Eating Disorder; Binge Eating
Keywords: Mobile Intervention; Adolescent
MeSH Terms: conditions — Obesity; Binge-Eating Disorder; Bulimia

STUDY DESIGN:
Intervention Model Description: Open trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Feasibility/Efficacy Testing Participants (Experimental): All participants will all be assigned to the experimental group in this single-arm open trial.
  Interventions: Behavioral: Feasibility/Efficacy Testing

INTERVENTIONS:
Behavioral: Feasibility/Efficacy Testing — This digital intervention will include elements of adapted cognitive-behavioral treatment for adolescent binge eating and weight control, with a focus on self-regulation and skills use.

SUMMARY:
The aim of this project is to pilot test a novel mobile app intervention for adolescents with dysregulated eating behaviors and elevated weight status. This intervention will incorporate evidence-informed strategies targeting self-regulation into cognitive-behavioral treatment for maladaptive eating. Adolescents will use the app for 16 weeks and provide feedback on its usability and effectiveness in managing dysregulated eating.

DETAILED DESCRIPTION:
This trial is part of a multi-phase project to create and test a mobile app intervention aimed at helping teenagers regulate their eating behaviors. Participation in this trial involves the following:

1. Adolescents and their parent are asked to attend a virtual assessment visit, where they will provide consent and complete questionnaires on eating-related thoughts and behaviors, mood, and experience with technology. The adolescent will also be asked to complete a semi-structured interview and provide height/weight measurements.
2. Eligible adolescents are then asked to complete a test-run week to make sure the trial is a good fit for them. They will be mailed a FitBit to wear continuously during the test-run week and a Smartscale to record their weight. They will also complete three 24-hour food recalls with a member of the research team during this week. Depending on engagement, the adolescent may or may not be invited to participate in the 16-week trial.
3. Adolescents eligible for the trial will use the VIBE app (Virtual Intervention for Binge Eating) and receive coaching for 16 weeks. Participants will also be asked to download an app that will help them with skill building and problem solving through short tasks/games, to be used while they are participating in the 16-week intervention.
4. Throughout the trial, adolescents will be invited to complete 3 additional assessment visits: "mid-point" or 8 weeks after starting the intervention, "post-intervention" at the end of the 16-week intervention, and "follow-up" 4 months after completing the intervention. These study assessments will include an interview, a weight measurement using the Smartscale, Fitbit usage for one week, up to 3 dietary recall phone calls, computerized tasks to assess how they think and solve problems, and online surveys. Each assessment will take about 90 - 120 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥75th percentile for their age and sex
* Report recent loss of control eating and/or overeating (≥3 episodes of either type of eating behavior in the past 3 months)
* Have an email address, Smartphone, and regular access to the internet
* Be willing and able to measure their height and weight prior to study enrollment

Exclusion Criteria:

* Report more than 2 instances of compensatory behavior (e.g. diuretics, laxatives, vomiting, driven exercise) in the past 3 months
* Not fluent in English at a third-grade reading level or higher
* Currently taking medications known to affect weight or appetite or concurrently involved in treatment for eating or weight disorders
* Meet criteria for a medical or psychiatric condition (e.g., diabetes, bulimia nervosa) known to significantly affect eating or weight, aside from binge eating disorder
* Developmental or cognitive delay precluding participation in the intervention
* Currently pregnant or lactating

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Usability of intervention | Week 16
  Perceptions that the intervention is or would be useful, useable, and satisfactory will be measured by the System Usability Scale.
Acceptability of intervention | Week 16
  Perceptions that the intervention is or would be useful, useable, and satisfactory will be measured by the Usefulness, Satisfaction, and Ease of use questionnaire (USE).
Body mass index percentile | Through study completion (up to 9 months)
  Adolescents will have their height and weight measured to calculate body mass index percentile using nationally representative growth charts and accompanying procedures. These data will be collected at each of the 4 major time points (pre-intervention assessment, mid-intervention assessment, post-intervention assessment, and 4-month follow up assessment).
Dysregulated eating | Through study completion (up to 9 months)
  Dysregulated eating (overeating and loss of control eating episodes) will be measured using the Eating Disorder Examination (EDE; interview and questionnaire). The EDE features 4 subscales that are rated on a 7-point forced-choice format (0-6), with higher scores reflecting greater severity or frequency. These measures will be completed at each of the 4 major time points (pre-intervention assessment, mid-intervention assessment, post-intervention assessment, and 4-month follow up assessment).

OTHER OUTCOMES:
Comorbid diagnoses | Pre-intervention assessment
  Comorbid psychiatric diagnoses will be reported by the adolescent's caregiver using the Child and Adolescent Symptom Inventory (CASI). Medical comorbid diagnoses will be reported by both the adolescent and their caregiver.
Intervention targets (activity patterns) | Through study completion (up to 9 months)
  Activity patterns (intervention target) will be measured using FitBit data during the intervention. Adolescents will track their activity using the FitBit over a 1-week period at each of the 4 major time points (pre-intervention assessment, mid-intervention assessment, post-intervention assessment, and 4-month follow up assessment).
Intervention targets (dietary patterns) | Through study completion (up to 9 months)
  Dietary patterns (intervention target) will be measured using phone-based 24-hour dietary recalls. Adolescents will complete 3 food recalls over a 1-week period at each of the 4 major time points (pre-intervention assessment, mid-intervention assessment, post-intervention assessment, and 4-month follow up assessment)
Putative treatment mechanisms (general) | Through study completion (up to 9 months)
  General self-regulation (putative mechanism) will be measured using the Self-Regulation Questionnaire. Items on the Self-Regulation Questionnaire are scored from 1 (strongly disagree) to 5 (strongly agree), with higher scores indicated higher self-regulation abilities. The questionnaire will be completed at each of the 4 major time points (pre-intervention assessment, mid-intervention assessment, post-intervention assessment, and 4-month follow up assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Goldschmidt, Ph.D., Principal Investigator — University of Pittsburgh; Andrea K Graham, Ph.D., Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Research data from participants may be shared with the broader scientific community after publication. We will make data and documentation available only under a data-sharing agreement that provides for a commitment to: (1) use the data for research purposes only; (2) secure the data using appropriate computer technology; (3) destroy or return the data after analyses are completed; and (4) not attempt to identify participants individually. Information shared with outside collaborators will link personal health information to a unique study ID in order to maintain participant anonymity.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Goldschmidt AB, Ortega A, Rooper IR, Obleada KT, Chapa DAN, Silverberg B, Stalvey E, Camino MK, Levine MD, Yu L, Eichen DM, Graham AK. Virtual Intervention for Binge Eating (VIBE): Study protocol for a user-informed mobile intervention for dysregulated eating and weight gain prevention in adolescents. Contemp Clin Trials. 2025 Dec 18;161:108192. doi: 10.1016/j.cct.2025.108192. Online ahead of print. PMID 41421758